CLINICAL TRIAL: NCT07162402
Title: Anxiety Among Children: Adaptation and Effectiveness of the Program Super Skills for Life in School Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatima Jinnah Women University (Other)
Responsible Party: Principal Investigator, Nazia Mustafa, Clinical Psychologist, Fatima Jinnah Women University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: FJWU/EC/2021/32
Record Dates: First submitted 2025-08-31; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Childhood Anxiety; Childhood Depression; Low Self-Esteem; Quality of Life (QOL); Social Skills; Emotional Problems; Behavioral Problems
Keywords: Anxiety and depressive symptoms, Pakistani Children, Super Skills for Life, Social skills, Quality of life
MeSH Terms: conditions — Social Skills; Problem Behavior; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: In the intervention arm, 8 sessions Super Skills for Life (SSL), were delivered to students who were screened positive for anxiety symptoms. Whereas Wait-list control group participants were not provided with intervention, they remained as usual with routine activities by teachers.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): In the intervention arm, 8 sessions Super Skills for Life (SSL), were delivered to students who were screened positive for anxiety symptoms
  Interventions: Other: Super Skills for Life (SSL) Program
- Wait-List Control Group (Other): Wait-list control group participants were not provided with intervention, they remained as usual with routine activities by teachers
  Interventions: Other: No Active Intervention

INTERVENTIONS:
Other: Super Skills for Life (SSL) Program — Its Cognitive Behaviour Therapy (CBT) Based 8 sessions Super Skills for Life (SSL) Program for childhood Anxiety Management.
  Arms: Intervention Group
Other: No Active Intervention — Routine Activities in Class
  Arms: Wait-List Control Group

SUMMARY:
Super Skills for Life (SSL) is a transdiagnostic prevention program designed for children with anxiety and depressive symptoms based on cognitive-behavioral therapy. This study is a Cluster Randomization Trial(cRCT) to determine the of the effectiveness of the SSL program to reduce anxiety and depressive symptoms along with improving self-esteem, social skills and overall quality of life in a sample of 126, 5th grade children recruited from 6 schools from Pakistan.

Schools were the unit of randomization and were randomly assigned to one of two experimental conditions; intervention group (SSL) and waiting list control (WLC) group. Assessments were conducted before and after the 8 sessions of intervention and follow-up assessment after 6 months.

DETAILED DESCRIPTION:
Super Skills for Life (SSL) is a transdiagnostic prevention program designed for children with anxiety and depressive symptoms based on cognitive-behavioral therapy. This study is a Cluster Randomization Trial(cRCT) to determine the of the effectiveness of the SSL program to reduce anxiety and depressive symptoms along with improving self-esteem, social skills and overall quality of life in a sample of 126, 5th grade children recruited from 6 schools from Pakistan.

Schools were the unit of randomization and were randomly assigned to one of two experimental conditions; intervention group (SSL) and waiting list control (WLC) group. Assessments were conducted before and after the 8 sessions of intervention and follow-up assessment after 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria of the study was a selection of children of Grade 5th presented with anxiety symptoms according to their scores equal to or greater than 25 on a total scale score of The Screen for Child Anxiety Related Emotional Disorders (SCARED) with age 9 and 13 years, who can speak and understand Urdu easily.

Exclusion Criteria:

* Children who have any serious physical/medical diseases, diagnosed mental health issues, developmental delays, or learning difficulties, and are under any psychological treatment were excluded. Furthermore, children who had undergone any surgery or experienced serious traumatic events in the past 6 months and who did not get permission from their parents with written informed consent from parents/ not willing to were also excluded.

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 126 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2021-09-16 (Actual); Study Completion 2021-09-16 (Actual)

PRIMARY OUTCOMES:
The Screen for Child Anxiety Related Emotional Disorders (SCARED) | Immediately after Intervention and Followup after 6 months
  Psychometric tool for Anxiety Measurement
The Center for Epidemiological Studies Depression Scale for Children (CES-DC) | Immediately post intervention and after 6 months
  Psychometric Tool for the measurement of Depression

SECONDARY OUTCOMES:
The Strength and Difficulties Questionnaire (SDQ) | Immediately post intervention and after 6 months
  Tool for the measurement of overall emotional and behavioural problems
Rosenberg Self-Esteem Scale (RSES) | Immediately after intervention and after 6 months
  Scale for assessing Self-Esteem
Social Skills Questionnaire (SSQ) | immediately after intervention and after 6 months
  tool for assessing Social Skills
Pediatric Quality of Life Inventory (PedsQL) | immediately after intervention and after 6 months
  tool for assessing Pediatric Quality of Life

CONTACTS AND LOCATIONS:
Locations (1):
- Fatima Jinnah Women University, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
will plan later after my publications